CLINICAL TRIAL: NCT02772146
Title: A Clinical Study of the Safety and Efficacy of a Wearable Device (CLS UF) That Delivers Continuous Administration of Glucose to Recirculated Peritoneal Dialysis Fluid for the Purpose of Ultrafiltration in Patients With Congestive Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After 2 patients it was concluded that a large change in exclusion criteria and study design was needed to obtain the ojective for the study
Sponsor: Triomed AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP Version 1D/2015-12-02; CIV-14-07-012440 (Other: Eudamed); Tmed-002 (Other: Triomed AB)
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure; Cardio-Renal Syndrome
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: CLS UF (Experimental): The purpose of CLS UF is ultrafiltration and drain of excess fluid in patients with congestive heart failure. The function of the device is to extra corporeally recirculate profiled glucose based PD fluid in a system and maintain glucose levels by adding extra glucose, to an adjustable and constant level, in order to maintain a stable ultrafiltration.
  Interventions: Device: CLS UF

INTERVENTIONS:
Device: CLS UF — One single ultrafiltration session of 10 hours.
  Other Names: Carry LifeTM System Ultra Filtration

SUMMARY:
A single-center, prospective, non-randomized, clinical and first-in-human study. Each patient will be studied during a single treatment session of ten hours. The device will be connected to an existing, standard PD catheter that the patient will be using routinely prior to the study (i.e. a peritoneal dialysis catheter will not be specifically inserted for the study). The patient will be hospitalized for observation during the test day and during the night following the study session. Ultrafiltration volume, dialysate glucose concentrations, blood glucose concentrations as well the patient's acceptability and tolerance of the wearable device will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, 18-80 years of age.
* Prevalent PD patients with CHF with cardio-renal syndrome type II, on stable ultrafiltration, for more than two months, treated with PD based UF according to German national guidelines.

  * Therapy resistance of pharmacologic therapy: resistant hypervolemia with ascites, pleural fluid and pulmonary edema
  * Recurrent hospitalization with cardiac decompensation, ≥ 2 occasions during the last six months
  * Isolated failure of the right heart chamber
* Treatment based on night time APD therapy combined with a day time long dwell.
* Obtained written consent to participate in the study.

Exclusion Criteria:

* End stage renal disease requiring dialysis.
* Malignant disease.
* On-going infection.
* Diabetes mellitus.
* HIV and/or hepatitis positive.
* Pregnancy.
* Breastfeeding women.
* Participation in other clinical trials within one month before inclusion.
* Abdominal hernia.
* Cardiac diseases other than left ventricular heart failure, biventricular heart failure or isolated right heart chamber failure, with volume overload.
* Any immune deficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Ultrafiltrated volume | 10 hours
  Ultrafiltrated volume during a 10 hours study session.

SECONDARY OUTCOMES:
Any Adverse Event (AE), Serious Adverse Event (SAE), Adverse Device Effect (ADE) or Serious Adverse Device Effect (SADE) occurring during the study session and until the follow-up visit. | 2-4 weeks
Patient acceptance of the wearable device | 10 hours
  Subjective opinion of each patient
Measured glucose levels in the re-circulated PD fluid | 10 hours
Patients acceptability of the re-circulation of PD fluid | 10 hours
  Any abdominal symptoms of the drain and fill of PD fluid will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Morath, PD Dr. Med, Principal Investigator — Division of Nephrology, Heidelberg University Hospital, Germany
Locations (1):
- Division of Nephrology, Heidelberg University Hospital, Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor may choose to publish or present data from this clinical investigation.